CLINICAL TRIAL: NCT06649279
Title: Variations in Oxygen Reserve Index in Different Fresh Gas Flow Rate
Brief Title: Oxygen Reserve Index in Different Fresh Gas Flow
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burak Kaya, Medical Doctor, Specialist, Sakarya University
Other Study IDs: E16214662-050.01.04-8172-213
Record Dates: First submitted 2024-10-11; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Oxygen Reserve Index
Keywords: Oxygen reserve index; Minimal flow anesthesia; High flow anesthesia; Hypoxia; Hyperoxia
MeSH Terms: conditions — Hypoxia; Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group H: High Flow Anesthesia Group
  Interventions: Device: Oxygen reserve index
- Group M: Minimal Flow Anesthesia Group
  Interventions: Device: Oxygen reserve index

INTERVENTIONS:
Device: Oxygen reserve index — Measuring oxygen reserve index during preoxygenation and under general anesthesia

SUMMARY:
Our primary objective is to determine whether oxygen reserve index ORI can be a reliable and sensitive indicator of hypoxia and hyperoxia in low-flow anesthesia settings. Our secondary objective is to investigate the ORI changes during preoxygenation stage.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* 18-75 years old
* underwent general anesthesia
* elective ear, nose and throat surgery, lasting longer than 60 minutes

Exclusion Criteria:

* who did not consent to participate,
* those with finger deformities
* unregulated diabetes mellitus, severe heart, kidney, or liver failure, sensitivities to local anesthetics or opioids, those who were morbidly obese (BMI >40 kg/m²), and breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective ear, nose, throat surgery.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Oxygen Reserve Index Value | For each patient, from preoxygenation stage to the end of the general anesthesia
  The Oxygen Reserve Index (ORI) is a real-time monitoring measure that captures the oxygen reserve status in the moderate hyperoxic range (PaO2 approximately 100 to 200 mmHg). ORI provides early warning of potential oxygenation disturbances before any changes occur in SpO2 and indicates the response to oxygen therapy. ORI ranges from 1 (high reserve) to 0 (no reserve) and measures changes in mixed venous oxygen saturation (SvO2) optically after arterial oxygen saturation reaches 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided